CLINICAL TRIAL: NCT07335497
Title: A Phase 1/2, Multicenter, Open-label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of CR-001 in Adult Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: CR-001 in Adult Participants With Locally Advanced or Metastatic Solid Tumors
Acronym: ASCEND
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Crescent Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR-001-101; 2025-523590-42-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced / Metastatic Solid Tumors
Keywords: solid tumors; metastatic; VEGF; PD-1; anti-PD-1; anti VEGF; immuno-oncology; anti-angiogenic therapy; checkpoint inhibitor; metastatic cancer; advanced cancer; First-in-Human; Dose Escalation; Dose Optimization
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CR-001 Dose escalation (Experimental): Escalating dose levels of CR-001 to define the maximum tolerated dose of CR-001 in participants with locally advanced or metastatic solid tumors who are refractory to or unable to tolerate standard of care treatment, or for whom standard of care treatment is unavailable
  Interventions: Drug: CR-001
- CR-001 Backfill (Experimental): Escalating dose levels of CR-001 Indication-specific cohort populations will be tested
  Interventions: Drug: CR-001
- CR-001 Dose Optimization Cohort X (Experimental): monotherapy dose level (DL)-X Indication-specific cohort populations will be tested
  Interventions: Drug: CR-001
- CR-001 Dose Optimization Cohort Y (Experimental): monotherapy DL-Y Indication-specific cohort populations will be tested
  Interventions: Drug: CR-001

INTERVENTIONS:
Drug: CR-001 — Intravenous Infusion

SUMMARY:
The purpose of this study is to determine the safety and tolerability of monotherapy CR-001 and identify the maximum tolerated dose (MTD), and/or optimal biologic dose and Recommended Phase 2 Dose(s) (RP2D) in participants with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The study will initially comprise 3 parts: dose escalation, backfill, and dose optimization cohorts. The study will follow a stepwise approach, beginning with a typical dose escalation in participants with selected indications of advanced solid tumors. Additional participants will enroll in the backfill part at select dose levels that have been previously cleared for safety by the safety review committee. In dose optimization, participants will be randomized to one of two CR-001 dose levels.

All participants will undergo a screening period, a treatment period of up to 2 years, a safety follow-up period, and long-term efficacy and survival follow-up. During the treatment period, participants will undergo clinical and safety assessments including disease assessment scans and blood laboratory safety, pharmacokinetic, and pharmacodynamic assessments. After treatment ends, disease scans will continue until disease progression, and long-term follow-up visits will be conducted by telephone every 3 months.

ELIGIBILITY:
Key Inclusion Criteria

* Life expectancy ≥ 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 - 1
* Adequate organ function and hematologic reserve based on laboratory parameters
* Have measurable disease defined by RECIST v1.1
* For Backfill and Dose Optimization: Willingness to provide recent archival tumor tissue sample or willingness to undergo biopsy
* Tumor Indication specific inclusion criteria:
* For dose escalation or backfill: progressing from, intolerant to, or ineligible for (due to unavailability or contraindication) local standard of care therapies and have one of the following locally advanced or metastatic tumor types:

  * Hepatocellular carcinoma
  * Biliary tract cancer
  * Endometrial carcinoma
  * Cervical cancer
  * Ovarian cancer
  * Gastric or gastroesophageal cancer
  * Colorectal cancer
  * Non-small cell lung cancer

Key Exclusion Criteria

* Has malignancies other than disease under study within the past 3 years
* Has conditions requiring treatment with clinically significant or increasing doses of systemic steroid therapy
* Has not adequately recovered from recent major surgery
* Has ongoing clinically significant toxicity related to prior therapy
* Has active central nervous system (CNS) metastases
* Has active autoimmune disease requiring systemic therapy in the past 2 years (replacement therapy is permitted)
* Has a history of serious Grade ≥ 3 immune-related adverse event (irAE)
* Has a history of noninfectious pneumonitis/interstitial lung disease
* Has an active severe infection
* Has received a live or attenuated vaccine within 30 days of the first dose
* Has undergone prior allogeneic stem cell or solid organ transplantation
* Has protocol-specified events related to gastrointestinal perforation, surgery, wound healing complications, and bleeding
* Has clinically significant cardiovascular disease NOTE: Other protocol defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation - Incidence and nature of dose-limiting toxicities | From the first dose of study drug up until approximately 1 month
  Per cohort
Dose Escalation - Characterization of the maximum tolerated dose, if applicable | From the first dose of study drug up until approximately 1 month
  Per Cohort
All parts - Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and treatment - emergent serious adverse events | From the first dose of study drug until 90 days after the last dose of study drug
  Events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
All parts - Incidence and severity of TEAEs leading to dose modifications | From the first dose of study drug until 90 days after the last dose of study drug
All parts - Incidence and severity of TEAEs leading to treatment discontinuation | From the first dose of study drug until 90 days after the last dose of study drug

SECONDARY OUTCOMES:
All parts - Determination of recommended Phase 2 dose(s) | From the first dose of study drug until 90 days after the last dose of study drug
All parts - Serum CR-001 pharmacokinetic parameters | Predose until up to approximately 36 months
  AUC0--inf after a single dose and steady state parameters, as appropriate
All parts - Serum CR-001 pharmacokinetic parameters | Predose until up to approximately 36 months
  AUClast after a single dose and steady state parameters, as appropriate
All parts - Serum CR-001 pharmacokinetic parameters | Predose until up to approximately 36 months
  Cmax after a single dose and steady state parameters, as appropriate
All parts - Serum CR-001 pharmacokinetic parameters | Predose until up to approximately 36 months
  Tmax after a single dose and steady state parameters, as appropriate
All parts - Serum CR-001 pharmacokinetic parameters | Predose until up to approximately 36 months
  Vd after a single dose and steady state parameters, as appropriate
All parts - Serum CR-001 pharmacokinetic parameters | Predose until up to approximately 36 months
  CL after a single dose and steady state parameters, as appropriate
All parts - Serum CR-001 pharmacokinetic parameters | Predose until up to approximately 36 months
  t½ after a single dose and steady state parameters, as appropriate
All parts - Incidence of participants with detectable antidrug antibodies | Predose until up to approximately 36 months
All parts - Overall response rate | From the first dose of study drug until up to approximately 36 months
All parts - Duration of response | From the first dose of study drug until up to approximately 36 months
All parts - Time to response | From the first dose of study drug until up to approximately 36 months
All parts - Progression free survival | From the first dose of study drug until up to approximately 36 months
All parts - Overall survival | From the first dose of study drug until up to approximately 36 months
All parts - Best percent change in target lesions | From the first dose of study drug until up to approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Brad Sumrow, MD, Study Director — Crescent Biopharma, Inc.
Locations (5):
- United States (5):
  - Clinical Study Site, Denver, Colorado
  - Clinical Study Site, Orlando, Florida
  - Clinical Study Site, Sarasota, Florida
  - Clinical Study Site, Nashville, Tennessee
  - Clinical Study Site, Dallas, Texas